CLINICAL TRIAL: NCT04444583
Title: Recognition of Heart Failure With Micro Electro-Mechanical Sensors (REFLECS) FI
Acronym: REFLECS-FI
Status: Completed | Type: Observational
Sponsor: Precordior Ltd (Industry)
Collaborators: Turku University Hospital (Other Government); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REFLECS-FI
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HFpEF: HF patients with preserved ejection fraction (HFpEF)
- HFrEF: HF patients with reduced ejection fraction (HFrEF)

SUMMARY:
In this study the ability of smartphone sensors (accelerometer and gyroscope) to identify patients with heart failure will be studied.

DETAILED DESCRIPTION:
Heart Failure (HF) is a condition where heart is unable to maintain adequate volume of blood in circulation corresponding to prevailing physiological demand. Gyrocardiography is a technique that utilizes micro electromechanical sensors (MEMS), accelerometer and gyroscope, to detect vibrations and rotation of thorax caused by cardiac motion. The main purpose of this study is to test the ability of an app of a smartphone with embedded motion sensors, positioned on the chest which measures the movements and function of the heart, to identify patients with different types of heart failure and their characteristics, as compared with clinical diagnosis. Echocardiography will also be used to confirm changes in cardiac cardiac mechanics including strain, cardiac torsion, diastolic filling characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients visiting hospital for heart failure, either outpatient clinic or cardiac ward
* Signed informed consent as an acceptance to participate to the trial

Exclusion Criteria:

* Age <18 years

  * Severe cardiac valve disease
  * Previous prosthetic cardiac valve
  * Major adverse cardiovascular event or surgery within 6 weeks of planned study enrollment
  * Patients with pacemaker
  * Informed consent form not signed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting Turku University Hospital Heart Center or Heart and Lung Center at Helsinki University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
HF specific motion sensor characteristics validation against echocardiography and other clinical features | From the hospital admission to study closure visit, on average 15 weeks
  The study aims to validate HF specific characteristics obtained with accelerometer (m/s2) and gyroscope (degree/s) against the current gold standard, detailed echocardiography examination in individuals already diagnosed with HF. Data of anonymised subjects without diagnosed or suspected HF will be used as controls to study the detection of HF.

SECONDARY OUTCOMES:
HF decompensation specific motion sensor characteristics validation | 14 weeks
  The ability of the motion sensors to detect differences in myocardial mechanics in patients with decompensation episode compared to patients without decompensation episode, assessed by receiver operating characteristics (ROC).

CONTACTS AND LOCATIONS:
Overall Officials: Antti Saraste, MD, PhD, Principal Investigator — Heart Center Turku University Hospital
Locations (2):
- Finland (2):
  - Heart and Lung Center at Helsinki University Hospital, Helsinki
  - Heart Center at Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No